CLINICAL TRIAL: NCT05809076
Title: Evaluation of the Effects of Gamma-tACS on the Periodic Activity of Neural Signals as a Function of State-dependency
Brief Title: Effects of Gamma-tACS on EEG Periodic Activity
Acronym: GAMMAtACS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS San Camillo, Venezia, Italy (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2021.18
Record Dates: First submitted 2023-03-16; First posted 2023-04-12 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-03

CONDITIONS: Transcranial Alternating Current Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- real tACS (Experimental)
  Interventions: Device: real tACS
- sham tACS (Sham Comparator)
  Interventions: Device: sham tACS

INTERVENTIONS:
Device: real tACS — tACS is a non-invasive method to induce brain modulation. It will be applied at a frequency of 40 Hz (gamma-tACS) with a peak-to-peak intensity of 2 mA. During the real tACS condition, the alternating current will be administered for 20 minutes.
  Arms: real tACS
Device: sham tACS — In the sham tACS condition, the current will be delivered only for the first 30 seconds and then stopped, in order to simulate the same somatosensory sensations as real tACS, but without inducing modulation.
  Arms: sham tACS

SUMMARY:
In this study on healthy subjects, the effect of transcranial alternating current stimulation (tACS) will be investigated. In particular, the distinction between periodic and aperiodic electroencephalogram (EEG) activity will be considered, as well as the state-dependency phenomenon. Participants will take part in two experimental sessions that will include tACS stimulation (one real, one control). Before, during, and after stimulation, subjects will have their EEG recorded during rest or during tasks.

The aim of this study is to investigate how the modulatory effects of gamma-tACS interact with intrinsic neural activity, measured in terms of periodic and aperiodic activity, as well as neurophysiological and behavioral modulation, taking into consideration the state-dependency phenomenon, which refers to the brain's activation state prior to stimulation.

ELIGIBILITY:
Inclusion Criteria:

- Healthy adults

Exclusion Criteria:

* Common exclusion criteria
* Left-handedness (assessed through the Oldfield test)
* Diagnosis of neurological or psychiatric disorders
* Vision problems that prevent reading, not correctable with lenses
* Diagnosis of substance dependence on drugs or alcohol
* Presence of hearing aids/prostheses
* Diagnosis of epilepsy or family history up to the second degree with it
* Episodes of febrile convulsions or recurrent fainting
* Head trauma
* Presence of surgical clips or metal implants in the head
* Diagnosis of heart disease
* Presence of a cardiac pacemaker or artificial heart valve
* Presence of hearing aids/prostheses
* Hearing problems or tinnitus
* Vision problems not corrected with lenses (such as color blindness)
* Taking tricyclic antidepressant medications
* Taking neuroleptic medications
* Diagnosis of headache or migraine
* Taking more than 3 alcoholic units in the last 24 hours
* Taking 2 or more cups of coffee or caffeine from other sources in the last 2 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2021-07-20 (Actual); Primary Completion 2023-01-18 (Actual); Study Completion 2023-01-18 (Actual)

PRIMARY OUTCOMES:
resting-state electroencephalography (EEG) signal | baseline
  The periodic and aperiodic activity of the EEG signal will be estimated through Brainstorm (i.e., EEG analysis software) and quantified in terms of numerical values representing the periodic/aperiodic component of the EEG signal. The periodic and aperiodic activity of the EEG signal will be assessed during three time frames: baseline, during the intervention, and immediately after the intervention (real or sham tACS)
resting-state electroencephalography (EEG) signal | during the intervension
  The periodic and aperiodic activity of the EEG signal will be estimated through Brainstorm (i.e., EEG analysis software) and quantified in terms of numerical values representing the periodic/aperiodic component of the EEG signal. The periodic and aperiodic activity of the EEG signal will be assessed during three time frames: baseline, during the intervention, and immediately after the intervention (real or sham tACS)
resting-state electroencephalography (EEG) signal | immediately after the intervention
  The periodic and aperiodic activity of the EEG signal will be estimated through Brainstorm (i.e., EEG analysis software) and quantified in terms of numerical values representing the periodic/aperiodic component of the EEG signal. The periodic and aperiodic activity of the EEG signal will be assessed during three time frames: baseline, during the intervention, and immediately after the intervention (real or sham tACS)

SECONDARY OUTCOMES:
behavioral performance (response times) | baseline
  Participants' motor performance at a computerized task will be measured in terms of response times (how fast the participants press a computer button, according to the task's instructions). The participants' motor performance will be assessed during two time frames: baseline and immediately after the intervention (real or sham tACS)
behavioral performance (response times) | immediately after the intervention
  Participants' motor performance at a computerized task will be measured in terms of response times (how fast the participants press a computer button, according to the task's instructions). The participants' motor performance will be assessed during two time frames: baseline and immediately after the intervention (real or sham tACS)
behavioral performance (accuracy) | baseline
  Participants' motor performance at a computerized task will be measured in terms of accuracy (% of correct responses at the computerized task, according to the task's instructions). The participants' motor performance will be assessed during two time frames: baseline and immediately after the intervention (real or sham tACS)
behavioral performance (accuracy) | immediately after the intervention
  Participants' motor performance at a computerized task will be measured in terms of accuracy (% of correct responses at the computerized task, according to the task's instructions). The participants' motor performance will be assessed during two time frames: baseline and immediately after the intervention (real or sham tACS)
auditory steady state response (ASSR) | baseline
  The auditory steady state response will be measured via EEG during entrainment through exposure to amplitude-modulated 40Hz sounds (5 min, sequence of amplitude-modulated tones at 40 Hz, delivered via earplug binaurally). The auditory steady state response will be measured as power of the EEG gamma band. The auditory steady state response will be assessed during two time frames: baseline and immediately after the intervention (real or sham tACS)
auditory steady state response (ASSR) | immediately after the intervention
  The auditory steady state response will be measured via EEG during entrainment through exposure to amplitude-modulated 40Hz sounds (5 min, sequence of amplitude-modulated tones at 40 Hz, delivered via earplug binaurally). The auditory steady state response will be measured as power of the EEG gamma band. The auditory steady state response will be assessed during two time frames: baseline and immediately after the intervention (real or sham tACS)

CONTACTS AND LOCATIONS:
Overall Officials: Arcara, Principal Investigator — IRCCS San Camillo Hospital
Locations (1):
- IRCCS San Camillo Hospital, Venice, Italy

IPD SHARING:
Plan to Share IPD: No